CLINICAL TRIAL: NCT04900350
Title: A Phase I/II Trial of AK117 (Anti-CD47) in Patients With Higher-risk Myelodysplastic Syndrome
Brief Title: A Trial of AK117 (Anti-CD47) in Patients With Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK117-103
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK117+ azacitidine (Experimental): Phase 1: Subjects will receive escalating doses of A117 in combination with azacitidine 75 mg/m2 subcutaneous daily for 7 days of a 28 day cycle;
  Phase 2: Subjects will receive AK117 at the recommended Phase 2 dose in combination with azacitidine 75 mg/m2 subcutaneous daily for 7 days of a 28-day cycle.
  Interventions: Drug: AK117; Drug: Azacitidine

INTERVENTIONS:
Drug: AK117 — Subjects receive AK117 intravenously.
Drug: Azacitidine — Subjects receive Azacitidine subcutaneously.

SUMMARY:
This is a open label, phase I/II study. All patients are diagnosed with higher-risk MDS, Eastern Cooperative Oncology Group (ECOG) performance status 0-2. The purpose of this study is to evaluate the safety and efficacy of AK117 + azacitidine in subjects with higher-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (at the time consent is obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Has a life expectancy of at least 12 weeks.
* Phase 1: Diagnosis of higher-risk MDS that is either previously untreated or relapsed/refractory.
* Phase 2: Diagnosis of higher-risk MDS that is previously untreated.
* White blood cell count ≤ 25 x 10^9/L (hydroxyurea may be used to reduce the WBC count).
* Has adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Is currently participating in a study of an investigational agent or using an investigational device.
* Has undergone major surgery within 30 days of Study Day 1.
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Previous allogeneic hematopoietic stem cell transplant (allo-HSCT) .
* Prior treatment with any anti-CD47 or anti-SIRPα (signal regulatory protein alpha) agent.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Remission (CR) | Approximately 6 months
  Number of participants achieving a CR per International Working Group (IWG) 2006 criteria.
Number of participants with adverse events (AEs) | Up to approximately 2 years.
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Duration of Complete Remission (DoCR) | Up to approximately 2 years.
  The DoCR is measured from the time measurement criteria are first met for CR to the first date of relapse or death, whichever occurs earlier.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years.
  ORR is defined as the proportion of participants who reach objective response including CR, Partial Remission (PR), marrow CR, or hematologic improvement per IWG 2006 MDS criteria prior to initiation of any new MDS therapy.
Duration of Response (DOR) | Up to approximately 2 years.
  DOR is measured from the time measurement criteria are first met for objective response to the first date of relapse or death, whichever occurs earlier.
Progression Free Survival (PFS) | Up to approximately 2 years.
  PFS is defined as the time from the start of treatment with AK117 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Maximum observed concentration (Cmax) of AK117 | Up to 2 years.
  Serum concentrations of AK117 in individual subjects at different time points after AK117 administration
Anti-drug antibodies (ADA) | Up to 2 years.
  Number of subjects with detectable anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China